CLINICAL TRIAL: NCT00206622
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study Comparing a 2.2mg 17 Beta-Estradiol/0.69mg Levonorgestrel Combination Transdermal Patch, and a 1mg 17 Beta-Estradiol Transdermal Patch With a Placebo Patch in Postmenopausal Women to Determine the Lowest Effective Dose of Estradiol for the Relief of Moderate to Severe Hot Flushes
Brief Title: Efficacy and Safety Study in Postmenopausal Women to Determine the Lowest Effective Dose for Relief of Moderate to Severe Hot-Flushes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91429; 308261
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — Estradiol

ARMS (3):
- Arm 1 (Active Comparator)
  Interventions: Drug: Climara PRO (Estradiol / Levonorgestrel transdermal)
- Arm 2 (Active Comparator)
  Interventions: Drug: Menostar (Estradiol transdermal)
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo transdermal

INTERVENTIONS:
Drug: Climara PRO (Estradiol / Levonorgestrel transdermal) — 2.2mg 17 Beta-estradiol/0.69mg levonorgestrel combination transdermal patch
  Arms: Arm 1
Drug: Menostar (Estradiol transdermal) — 1mg 17 Beta-estradiol transdermal patch
  Arms: Arm 2
Drug: Placebo transdermal — Placebo
  Arms: Arm 3

SUMMARY:
To determine the lowest effective dose of estradiol by comparing E2/LNG (2.2mg/0.69mg) and E2 (1.0mg) dose with placebo in decreasing the frequency and severity of moderate to severe hot flushes in postmenopausal women

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.

Bayer HealthCare Pharmaceuticals, Inc.is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Menopause
* Reporting a minimum of 7 moderate to severe hot flushes per day for at least 1 week (7 consecutive days), or a minimum of 50 moderate to severe hot flushes per week for at least 1 week (7 consecutive days)

Exclusion Criteria:

* Hormonal treatment
* Contraindication to estrogen/progestogen therapy

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2004-12; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Lowest effective dose in decreasing the frequency and severity of hot flushes

SECONDARY OUTCOMES:
Other symptoms related to menopause

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (41):
- United States (41):
  - Huntsville, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Fair Oaks, California
  - Oakland, California
  - San Diego, California
  - New Britain, Connecticut
  - West Hartford, Connecticut
  - Fort Myers, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Alpharetta, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Champaign, Illinois
  - Chicago, Illinois
  - Peoria, Illinois
  - South Bend, Indiana
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Detroit, Michigan
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Reno, Nevada
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Memphis, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - Temple, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont

REFERENCES:
- [Derived] Bachmann GA, Schaefers M, Uddin A, Utian WH. Lowest effective transdermal 17beta-estradiol dose for relief of hot flushes in postmenopausal women: a randomized controlled trial. Obstet Gynecol. 2007 Oct;110(4):771-9. doi: 10.1097/01.AOG.0000284450.51264.31. PMID 17906008